CLINICAL TRIAL: NCT01790516
Title: A Pilot Prospective Clinical Trial to Use Pharmacogenetics (PGx) to Select Erbitux or Cisplatin to Treat Head and Neck Cancer
Brief Title: Use of Pharmacogenetics to Select Erbitux or Cisplatin to Treat Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accruals--2 patients were enrolled in over a year
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-439
Record Dates: First submitted 2012-06-21; First posted 2013-02-13 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2013-10

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: Head and neck cancer; genetic testing; cisplatin; erbitux; radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Platinum; Cetuximab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin (Experimental): Cisplatin
  Interventions: Drug: Cisplatin; Radiation: Radiation
- Cetuximab (Experimental): cetuximab
  Interventions: Drug: cetuximab; Radiation: Radiation

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 100 mg/m2 during weeks 1,4, and 7 of radiation therapy
  Other Names: Cispaltin; Platinum
  Arms: Cisplatin
Drug: cetuximab — Cetuximab beginning at a dose of 400 mg/m2 the week before radiation commences and then 250 mg/m2 weekly during weeks 1 and 7 of radiation.
  Other Names: Erbitux
  Arms: Cetuximab
Radiation: Radiation — daily radiation for 7 weeks

SUMMARY:
This study is for patients with newly diagnosed head and neck cancer that cannot be removed by surgery.

The purpose of this study is to determine the feasibility of using genetic variations in patients to select the right drug to treat head and neck cancer. Cisplatin and cetuximab (Erbitux)are both approved by the FDA to treat head and neck cancer in combination with radiation therapy. In this study the investigators will test whether genetic differences between patients can be used to pick which of these two drugs a patient should receive. All patients will have a blood sample drawn that will be tested for genetic differences. If patients have genetic differences that correlate with a better outcome from cisplatin they will receive cisplatin with radiation. If patients have genetic differences that do not correlate with a better outcome from cisplatin they will receive cetuximab with their radiation therapy.

DETAILED DESCRIPTION:
Treatment-naive patients with locally advanced, non-metastatic (Stage III to IVB) squamous cell carcinoma of the head and neck who are candidates for concurrent chemoradiotherapy as primary therapy with curative intent will be enrolled. Patients will be genotyped for germline variations at four SNP loci in three genes involved in DNA nucleotide excision repair (ERCC1, ERCC2, and XRCC1). Patients with 3 to 8 variants will receive cisplatin (Arm A). Patients with 2 or fewer variants will receive cetuximab (Arm B).

The hypothesis of the study is that prospectively testing patients for variations in DNA repair enzymes to determine whether to use cisplatin or cetuximab in locally advanced head and neck squamous cell cancer is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the head and neck, including the oral cavity, oropharynx, hypopharynx, or larynx, but not including primary tumors of the nasopharynx, sinuses, or salivary glands.
* Locally advanced, Stage III to IVB disease, and a candidate for primary therapy using chemotherapy and radiation therapy with curative intent.
* Patients with a diagnosis of 'unknown primary' will be eligible if chemoradiotherapy is the primary modality of treatment
* No previous chemotherapy, radiation, or surgery for their diagnosis of head and neck cancer
* Eastern Cooperative Oncology Group performance status </= 1
* Women of child-bearing potential must have a negative pregnancy test within 30 hours before initiation of study drug dosing. Female subjects of reproductive potential must agree to avoid pregnancy throughout the study and for up to 3 months following discontinuation of study drug. Male subjects must agree to avoid conceiving a child throughout the study and for up to 3 months following discontinuation of study drug;
* Hemoglobin >/= 8.0 gm/dL
* Absolute neutrophil count >/= 1500
* Platelet count >/= 100,000
* Glomerular Filtration Rate > 50 mL/min calculated by the Cockcroft-Gault equation
* Total bilirubin </= 2.0 times the upper limit of normal unless the patient has Gilbert's syndrome
* Aspartate aminotransferase and Alanine Aminotransferase </= 2.5 times the upper limit of normal
* No other current malignancy, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular in situ of the breast. Patients with other malignancies are eligible if they have been continuously disease-free for >/= 3 years prior to screening for this protocol.
* Age of 18 or older
* Ability and willingness to give informed consent
* Subjects must in the opinion of the Investigator be capable of complying with this protocol.

Exclusion Criteria:

* Acute treatment for an infection or other serious medical illness within 14 days prior to study entry
* Major surgery within 3 weeks prior to study entry
* Known hypersensitivity to cisplatin or cetuximab
* Patients who have any severe or uncontrolled medical conditions or other conditions that could affect their participation in this study, including: unstable angina, serious uncontrolled cardiac arrhythmia, active acute or uncontrolled infectious disorder, or myocardial infarction </= 6 months prior to study entry.
* Female patients who are pregnant or breast feeding, or adults who are of reproductive potential and are unwilling to refrain from conceiving a child during study treatment.
* Patients unwilling to comply with the protocol, or provide informed consent
* Psychiatric illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Deeken, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprhensive Cancer Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin: Intensity modulated radiation with concurrent cisplatin
  platinum plus radiation: Cisplatin 100 mg/m2 during weeks 1,4, and 7 of radiation therapy
- Cetuximab: Intensity modulated radiation therapy with concurrent cetuximab
  cetuximab plus radiation therapy: Cetuximab beginning at a dose of 400 mg/m2 the week before radiation commences and then 250 mg/m2 weekly during weeks 1 and 7 of radiation.
Period: Overall Study
Arm/Group | Cisplatin | Cetuximab
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: male, caucasian, adult over 18
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin | Cetuximab | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Returning Genetic Testing Results in a Timely Manner to the Treating Physician
Description: Feasibility is defined as follows:
  - Patients' genetic test results are returned to the treating physician within 3 days
Time Frame: 20 months
Measure: Median (Full Range); unit: days
Arm/Group | Cisplatin | Cetuximab
Number analyzed (Participants) | 1 | 1
days | 3 [3 to 3] | 3 [3 to 3]

ADVERSE EVENTS:
Arm/Group | Cisplatin | Cetuximab
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No